CLINICAL TRIAL: NCT04295759
Title: A Phase I Study of the Adam-10 Inhibitor, INCB7839 in Children With Recurrent/Progressive High-Grade Gliomas to Target Microenvironmental Neuroligin-3
Brief Title: INCB7839 in Treating Children With Recurrent/Progressive High-Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); American Lebanese Syrian Associated Charities (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-056; UM1CA081457 (NIH); PBTC-056 (Other: Pediatric Brain Tumor Consortium); PBTC-056 (Other: CTEP); NCI-2019-08964 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-02-27; First posted 2020-03-04 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; DIPG; High-grade Astrocytoma NOS; CNS Primary Tumor, NOS (Malignant Glioma)
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Pyloric Stenosis, Hypertrophic; Glioma

STUDY DESIGN:
Intervention Model Description: This is a phase I study and we will use a design similar to the Rolling-6 design and open 6 slots initially on Dose level 1. If we observe no-more than 1 DLT in these 6 subjects then we would expand this cohort to at least 12 patients for PK and additional safety information. If more than 1 DLT is observed on dose level 1 in 2-6 subjects, then further enrollment to dose level 1 will stop, the dose will be de-escalated to dose level 0 and the same approach will be repeated. Based on the above-outlined de-escalation rules, if dose level 0 is found to be too toxic, then the trial will be closed to accrual and the merits of amending or closing the trial permanently will be reconsidered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose-finding (Experimental): INCB7839 dosing will begin at 120 mg/m2/dose BID which is equivalent to the adult RP2D (200 mg PO BID) based on a typical adult size of 1.67m2. The INCB7839 dose may be decreased to 80 mg/m2/dose BID if the staring dose is not tolerable. 28 consecutive days (4 weeks) will constitute one course. Patients may continue to receive INCB7839 for 26 courses (approximately 2 years).
  Interventions: Drug: INCB7839

INTERVENTIONS:
Drug: INCB7839 — INCB7839 dosing will begin at 120 mg/m2/dose BID which is equivalent to the adult RP2D (200 mg PO BID) based on a typical adult size of 1.67m2. The INCB7839 dose may be decreased to 80 mg/m2/dose BID if the staring dose is not tolerable. 28 consecutive days (4 weeks) will constitute one course. Patients may continue to receive INCB7839 for 26 courses (approximately 2 years).

SUMMARY:
This is a multicenter phase 1 trial of INCB7839 for children with recurrent or progressive high-grade gliomas, including, but not limited to, diffuse intrinsic pontine glioma (DIPG) and other diffuse midline gliomas (DMGs), after upfront therapy.

DETAILED DESCRIPTION:
INCB7839 is an inhibitor of the ADAM (A Disintegrin and Metalloprotease) 10 and 17 proteases. Neuronal activity regulates glioma growth through neuroligin-3 (NLGN3). ADAM 10 is the protease responsible for NLGN3 release into the tumor microenvironment and represents a promising therapeutic target.

Pre-clinical studies of INCB7839 in patient-derived pediatric high-grade gliomas (GBM and DIPG) revealed that INCB7839 inhibits pediatric high- grade glioma growth and improves overall survival. In vivo testing also demonstrated that INCB7839 penetrates brain tissue sufficient to achieve its pharmacodynamic effect of ADAM10 inhibition. Further pre-clinical studies in other animals revealed minimal toxicity, including non-adverse to mild increases in serum hepatobiliary enzymes, protein, calcium, cholesterol values, along with minimal decreases in RBC mass parameters; all parameters recovered.

INCB7839 has been evaluated in Phase I and Phase II clinical trials for previously treated solid tumors and breast cancer. Of the adverse events (AEs) noted, the majority were mild-to-moderate in severity, the most frequent being fatigue, nausea, anorexia, diarrhea, emesis, abdominal pain, anemia and constipation. The dose-limiting toxicity for monotherapy with INCB7839 in Phase I clinical trials was declared to be deep venous thrombosis (DVT). Out of 41 patients, there was a total of 9 thrombotic events including mild superficial thrombophlebitis (n=1), DVT (n=4), vena cava thrombosis with renal insufficiency in a patient with squamous cell cancer of the head and neck (n=1), atrial thrombosis in patient with breast cancer (n=1), and pulmonary embolism in patients with hormone-refractory prostate cancer (n=2). Overall, INCB7839 does exhibit a pro-coagulant effect in some adult patients, resulting in an increased incidence of DVT, whether used alone or in combination. The mechanism of this effect is unknown, and there is no clear relationship between the frequency of thrombosis and the dose administered.

ELIGIBILITY:
INCLUSION CRITERIA:

Histologic diagnosis:

* Patients with recurrent/progressive high-grade gliomas, as defined by progressive neurologic abnormalities or worsening neurologic status not explained by causes unrelated to tumor progression (e.g., anticonvulsant or corticosteroid wean, electrolyte disturbances, sepsis, hyperglycemia, etc.), OR a ≥ 25% increase in the bi-dimensional measurement, taking as a reference the smallest disease measurement recorded since diagnosis utilizing the MRI sequence best demonstrating tumor, OR the appearance of a new/metastatic tumor lesion(s) since diagnosis.
* Eligible diagnoses include but are not limited to the following: diffuse intrinsic pontine glioma (DIPG), H3K27M-altered diffuse midline glioma (DMG), glioblastoma multiforme, anaplastic astrocytoma and anaplastic oligodendroglioma. Spinal cord tumors are eligible with pathologic confirmation of the above.
* Please note: Patients with a radiographically typical DIPG at diagnosis, defined as a tumor with a pontine epicenter and diffuse involvement of more than 2/3 of the pons, are eligible without histologic confirmation.
* Patients with pontine lesions that do not meet these radiographic criteria will be eligible if there is histologic confirmation of pontine glioma WHO II-IV.
* Patients with diffuse or multi-focal disease are eligible; patients with leptomeningeal spread are eligible.

Age

* Patients must be ≥ 3 but ≤ 21 years of age at the time of enrollment.

BSA

* Patients must have a BSA ≥ 0.70-2.50 m2 for dose 120 mg/m2/dose BID.
* Patients must have a BSA ≥ 0.55-2.80 m2 for dose 80 mg/m2/dose BID (Patients who have BSA 0.55-1.00 m2 will only receive 100 mg AM dose).

Ability to Swallow

* Patients must be able to swallow tablets whole.

Measurable disease

* Patients must have measurable disease in two dimensions on MRI to be eligible.

Prior Therapy

* Patients must have failed at least 1 standard, tumor-directed treatment besides surgery and recovered from the acute treatment-related toxicities (defined as < Grade 1) of all prior chemotherapy, immunotherapy, or radiotherapy prior to enrollment on this study.
* Patients must be ≥ 28 days from any prior surgery at the time of study enrollment (with the exception of minor dental and dermatological procedures).

  * Chemotherapy
* Patients must have received their last dose of known myelosuppressive anticancer therapy at least 21 days prior to enrollment or at least 42 days if nitrosourea.

  * Investigational/ Biologic Agent
* Biologic or investigational agent (anti-neoplastic): Patients must have recovered from any acute toxicity potentially related to the agent and received their last dose of the investigational or biologic agent ≥ 7 days prior to study enrollment.
* For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
* Monoclonal antibody treatment and agents with known prolonged half-lives: Patients must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 28 days prior to study enrollment.
* Immunotherapies: Patients who have received checkpoint inhibitors or other immunotherapies with a known potential for pseudoprogression and who have assumed tumor progression must be at least 12 weeks from prior immunotherapy AND have at least two MRI scans at least 4 weeks apart demonstrating further progression OR have a biopsy to confirm tumor progression OR have new site(s) of disease.

  * Radiation

Patients must have had their last fraction of:

* Craniospinal irradiation, whole brain radiation, total body irradiation or radiation to ≥ 50% of pelvis or spine ≥ 42 days prior to enrollment.
* Focal irradiation ≥ 14 days prior to enrollment.
* Local palliative irradiation to site other than primary tumor progression site ≥ 14 days prior to enrollment.
* Stem Cell Transplant

Patients must be:

* ≥ 6 months since allogeneic stem cell transplant prior to enrollment with no evidence of active graft vs. host disease.
* ≥ 3 months since autologous stem cell transplant prior to enrollment.

Neurologic Status

* Patients with neurological deficits should have deficits that are stable for a minimum of 7 days prior to enrollment.
* Patients with seizure disorders may be enrolled if seizures are well controlled.

Performance Status

* Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) assessed within two weeks of enrollment must be ≥ 50.

Organ Function: Patients must have adequate organ and marrow function as defined below:

* Absolute neutrophil count ≥ 1.0 x 10^9 cells/ L
* Platelets > 100 x 10^9 cells/ L (unsupported, defined as no platelet transfusion within 7 days)
* Hemoglobin ≥ 8 g/dL (may receive transfusions)
* Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN)
* ALT (SGPT) and AST (SGOT) < 3 x institutional upper limit of normal (ULN)
* Albumin ≥ 2 g/dL
* Serum creatinine based on age/gender as noted in institutional normal range. Patients that are not within institutional normal range but have a 24-hour Creatinine Clearance or GFR (radioisotope or iothalamate) ≥ 70 mL/min/1.73 m^2 are eligible.

Corticosteroids

* Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 7 days prior to enrollment.

Growth Factors

* Patients must be off all colony-forming growth factor(s) for at least 7 days prior to enrollment (e.g., filgrastim, sargramostim or erythropoietin). Fourteen (14) days must have elapsed if patient received a long-acting formulation.

Pregnancy Prevention

* Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.

Informed Consent

* The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document according to institutional guidelines.

HIV Positive Patients

* HIV-positive patients are eligible if the following criteria are met:

  * Stable on their antiretroviral agents
  * Have CD4 counts above 400/mm^3
  * Undetectable viral loads, and
  * No need for prophylactic medications for an opportunistic infections

EXCLUSION CRITERIA:

Pregnancy or Breast-feeding

* Pregnant women or nursing mothers are excluded from this study. Female patients of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  * Pregnant or breast-feeding women are excluded from this study due to risks of fetal and teratogenic adverse events as seen in animal studies.

Concurrent Illness

* Patients with any clinically significant unrelated systemic illness (e.g., serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results.
* Patients with any other current malignancy.
* Patients with uncontrolled hypertension (i.e., a blood pressure (BP) > 95th percentile for age, height, and gender; patients with values above these levels must have their blood pressure controlled with medication prior to starting study drug).

  * The normal blood pressure by height, age, and gender tables can be accessed in the Generic Forms section of the PBTC member's webpage.
  * Patients who are ≥ 18 years of age must have blood pressure that is < 140/90 mm of Hg at the time of registration.

Concomitant Medications

* Patients who are receiving any other anti-cancer, investigational or alternative (e.g., cannabinoids) drug therapy are ineligible.

Prisoners

* Prisoners will be excluded from this study.

Inability to participate

* Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures and study restrictions.

Allergy

* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition.
* Patients with a history of allergy to pork products due to contraindications with low molecular weight heparin (LMWH).

Thrombosis Risk

* Patients with a known coagulopathy or bleeding disorder (e.g., von Willebrands disease) are not eligible.
* Patients with a history of non-central line related thrombosis or disorders that promote clotting (e.g., anti-thrombin III deficiency, Lupus anticoagulant) are not eligible.
* Significant family history of thrombosis (i.e. deep venous thrombosis or pulmonary embolus) in a first-degree relatives (i.e., parents or siblings) are not eligible.
* Estrogen containing contraceptives are not permitted due to thrombotic risk. Progestin-only contraception along with alternate forms of contraception are acceptable.
* Patients should be counseled to avoid smoking/tobacco products.
* If there is any contraindication to DVT prophylaxis, the patient is not eligible.

Family history must be documented to the best extent it is known.

Subjects with current or prior symptomatic intratumoral or intracranial hemorrhage are ineligible.

Subjects with asymptomatic evidence of new CNS hemorrhage of more than punctate size (i.e., ≥ 4 mm) and/or more than one punctate focus of hemorrhage (< 4 mm or not seen on more than one slice) on baseline MRI obtained within 14 days prior to study enrollment are ineligible.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Monje, MD, PhD, Study Chair — Stanford University and Lucile Packard Children's Hospital
Locations (11):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University and Lucile Packard Children's Hospital, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children Hospital Medical Center, Cincinnati, Ohio
  - Children Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients ≥3 and ≤21 years of age with recurrent or progressive high-grade gliomas including but not limited to diffuse intrinsic pontine glioma (DIPG) and other diffuse high-grade gliomas were enrolled at Pediatric Brain Tumor Consortium (PBTC) member institutions. The first patient was enrolled on 7/27/2020 and the last patient was enrolled on 2/7/2023. Only one dose level was studied; all subjects were enrolled on Dose Level 1 (120 mg/m^2/dose).
Groups:
- Dose Level 1 (120 mg/m^2/Dose): Subjects with recurrent or progressive high-grade gliomas received 120 mg/m^2/dose of INCB7839 orally, twice a day for 28-day cycles. Treatment could continue for up to 26 courses (approximately 2 years) in the absence of disease progression or unacceptable toxicity or another off treatment or off study reason.
Period: Overall Study
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Started | 13
Completed | 0
Not Completed | 13
Not completed — Lack of Efficacy | 9
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Deemed ineligible | 1

BASELINE CHARACTERISTICS:
Population: Summary statistics for baseline characteristics are shown for eligible patients only (n=12). One subject was deemed ineligible. All subjects received Dose Level 1.
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 14.5 [4.9 to 20.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced Dose-limiting Toxicities (DLTs)
Description: All subjects evaluable for dose-finding were classified as having DLT or not having DLT, and the number of subjects having DLT was reported. Any INCB7839-related adverse events during the first course of treatment that led to dose reduction, permanent cessation of therapy, or a delay in treatment of >7 days were considered DLTs. Hematologic DLTs included any grade 4 hematologic toxicity except lymphopenia; grade 3 neutropenia with fever; or requiring a platelet transfusion on 2 separate days during a single course. Non-hematologic DLTs included any grade 4 non-hematologic toxicity; any grade 3 non-hematologic toxicities with some exceptions such as grade 3 fever or infection of fewer than 5 days in duration; any grade 2 non-hematologic toxicity persisting for >7 days and considered medically significant; and any deep venous thrombotic event (superficial phlebitis was excluded unless grade 3 or 4 or unless it met another criteria for DLT).
Time Frame: Approximately 28 days
Population: Only eligible subjects and those evaluable for estimating the maximum tolerated dose (MTD) were included in this analysis (n=10). Of 13 subjects enrolled, 1 was deemed ineligible, and 2 were not evaluable for dose-finding as they received less than 85% of planned INCB7839 dosing during the dose-finding period for reasons other than toxicity, including 1 subject who withdrew prior to beginning therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 10
Participants | 3

2. Primary Outcome: Maximum Tolerated Dose (MTD) and/or Recommend Phase II Dose (RP2D) of INCB7839
Description: A design similar to the Rolling-6 design was used and 6 slots were initially opened on the starting dose level (dose level 1, INCB7839 120 mg/m^2/dose BID). If no more than one dose-limiting toxicity (DLT) was observed in these 6 subjects, we would expand this cohort to at least 12 patients for additional safety and pharmacokinetic information. If more than 3 DLTs were observed in 12 subjects at dose level 1, then the initially identified maximum tolerated dose based on 6 subjects would be considered unsafe and de-escalation to a lower dose level (INCB7839 80 mg/m^2/dose BID) would be considered.
Time Frame: Approximately 28 days
Population: Of 13 subjects enrolled, 1 was deemed ineligible, and 2 were not evaluable for dose-finding as they received less than 85% of planned INCB7839 dosing during the dose-finding period for reasons other than toxicity, including 1 subject who withdrew prior to beginning therapy. Because we had 10 eligible, evaluable subjects rather than the required 12 needed to address this objective, we were unable to define the MTD and no result is reported.
Measure: Number; unit: mg/m^2/dose
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 10
mg/m^2/dose | NA — Because we had 10 eligible, evaluable subjects rather than the required 12 needed to address this objective, we were unable to define the MTD and no result is available or reported for this outcome measure.

3. Primary Outcome: Area Under the Curve (AUC) of INCB7839
Description: Pharmacokinetic (PK) studies were performed after an oral INCB7839 dose on days 1, 2, and 3 of Course 1. Beginning day 1 of Course 1, INCB7839 serial blood PK samples were drawn pre-dose and at approximately 1, 4, 8, 24, and 48 hours after the first dose. Time points at which data were collected to create the curve were 0, 1, 4, 8, 24 and 48 hours post-dose. The area under the curve (AUC) was estimated using a noncompartmental method.
Time Frame: Up to 3 days after the start of treatment
Population: Eligible patients who had PK samples collected and had AUC data available were included in this analysis.
Measure: Median (Full Range); unit: h*ng/ml
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 11
h*ng/ml | 3852 [1820 to 8638]

4. Primary Outcome: Maximum Concentration [Cmax] of INCB7839
Description: Pharmacokinetic (PK) studies were performed after an oral INCB7839 dose on days 1, 2, and 3 of Course 1. Beginning day 1 of Course 1, INCB7839 serial blood PK samples were drawn pre-dose and at approximately 1, 4, 8, 24, and 48 hours after the first dose. Time points at which data were collected were 0, 1, 4, 8, 24 and 48 hours post-dose. The maximum concentration (Cmax) was estimated using a noncompartmental method.
Time Frame: Up to 3 days after the start of treatment
Population: Eligible patients who had PK samples collected and who had Cmax data available were included.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 11
ng/ml | 558 [130 to 1262]

5. Primary Outcome: Apparent Oral Clearance [CL/F] of INCB7839
Description: Pharmacokinetic (PK) studies were performed after an oral INCB7839 dose on days 1, 2, and 3 of Course 1. Beginning day 1 of Course 1, INCB7839 serial blood PK samples were drawn pre-dose and at approximately 1, 4, 8, 24, and 48 hours after the first dose. Time points at which data were collected were 0, 1, 4, 8, 24 and 48 hours post-dose. Clearance (CL/F) was estimated using a noncompartmental method.
Time Frame: Up to 3 days after the start of treatment
Population: Eligible patients who had PK samples collected and who had CL/F data available were included.
Measure: Median (Full Range); unit: L/hr/m^2
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 11
L/hr/m^2 | 34.6 [18.5 to 68.5]

6. Primary Outcome: Time to Reach Maximum Concentration [Tmax] of INCB7839
Description: Pharmacokinetic (PK) studies were performed after an oral INCB7839 dose on days 1, 2, and 3 of Course 1. Beginning day 1 of Course 1, INCB7839 serial blood PK samples were drawn pre-dose and at approximately 1, 4, 8, 24, and 48 hours after the first dose. Time points at which data were collected were 0, 1, 4, 8, 24 and 48 hours post-dose. The time to reach maximum concentration (Tmax) was estimated using a noncompartmental method.
Time Frame: Up to 3 days after the start of treatment
Population: Eligible patients who had PK samples collected and who had Tmax data available were included.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 11
hours | 4.0 [3.9 to 8.4]

7. Secondary Outcome: Percent Probability of Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time interval from date of treatment start to date of first event (progressive disease or death due to any cause) for patients with events, or to the date of last follow-up for patients without events. PFS was estimated using the method of Kaplan and Meier and reported with a 95% confidence interval. We had planned to report the 2-year PFS estimate, but the 2-year estimate was not defined as most subjects progressed prior to 2 years. The 3-month PFS estimate was reported. All subjects are off study and data collection has concluded for this outcome measure.
Time Frame: 3 months from first dose of INCB7839
Population: Of 12 eligible subjects enrolled, 1 did not start therapy and therefore was not evaluable for efficacy evaluation and estimation of PFS.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 11
Percent probability | 18.18 [0 to 40.97]

8. Secondary Outcome: Percent Probability of Overall Survival
Description: Overall survival (OS) was defined as the time interval from date of treatment initiation to date of death due to any cause or to the date of last follow-up for survivors. OS was estimated using the method of Kaplan and Meier and reported with a 95% confidence interval. All subjects are off study and data collection has concluded for this outcome measure.
Time Frame: 3 months from first dose of INCB7839
Population: Of 12 eligible subjects enrolled, 1 did not start therapy and therefore was not evaluable for efficacy evaluation and estimation of overall survival.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 11
Percent probability | 53.69 [17.02 to 90.36]

9. Secondary Outcome: Duration of Response
Description: Complete or partial responses were considered responses. Response was evaluated by imaging or clinical progression. Duration of response was measured from the time measurement criteria were met for complete or partial response until the first date that recurrent or progressive disease was objectively documented.
Time Frame: Up to 2 years following last dose of INCB7839
Population: Of 12 eligible subjects enrolled, 1 did not start therapy and therefore was not evaluable for response. Among 11 eligible, evaluable subjects, none had complete or partial responses, and it was not possible to calculate duration of response.
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: ADAM10 Inhibition of HER2
Description: HER2 extracellular domain (ECD) in serum will be reported.
Time Frame: Baseline and Day 14 of Course 1
Population: Eligible subjects with HER2 ECD data were included in this analysis. Ten participants had data at baseline and 9 had data at day 14 of course 1.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 10
ng/ml
  Baseline | 16.66 [4.24 to 37.26]
  Course 1, Day 14 | 17.55 [4.64 to 114.00]

11. Other Pre Specified Outcome: ADAM10 Inhibition of Neuroligin-3 (NLGN3)
Description: Descriptive statistics for neuroligin-3 (NLGN3) in cerebral spinal fluid will be reported.
Time Frame: Up to 30 days post treatment.
Population: No samples were received for this exploratory objective.
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Maximum Concentration [CMAX] of INCB7839 in Cerebrospinal Fluid
Description: The maximum concentration [CMAX] will be calculated based on the cerebrospinal fluid pharmacokinetic samples.
Time Frame: Up to 30 days post treatment
Population: No samples were received for this exploratory objective.
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected while participants were on protocol therapy and up to 6 months while in follow-up
Description: Only eligible subjects that started therapy were included in adverse event (AE) reporting (n=11). As per protocol, grade 1-2 AEs that were at least possibly related to drug and all grade 3-5 AEs regardless of attribution to study drug were recorded. AEs were graded using CTCAE v5.0. Serious AEs included those that were life-threatening or AEs requiring intervention, resulting in death, hospitalization, disability, congenital anomaly/birth defect or otherwise marked serious in Rave.
Arm/Group | Dose Level 1 (120 mg/m^2/Dose)
All-Cause Mortality (participants affected / at risk) | 4/11
Serious Adverse Events (participants affected / at risk) | 9/11
Other Adverse Events (participants affected / at risk) | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (120 mg/m^2/Dose) (N=11)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Death NOS (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cerebral Venous Thrombosis (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hydrocephalus (Nervous system disorders) | 4 (4)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Paroxysmal Sympathetic Hyperactivity (Nervous system disorders) | 1 (1)
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (3)
Somnolence (Nervous system disorders) | 2 (2)
Spasticity (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (120 mg/m^2/Dose) (N=11)
Anemia (Blood and lymphatic system disorders) | 3 (10)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (6)
Fever (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (13)
Aspartate aminotransferase increased (Investigations) | 4 (6)
Hemoglobin increased (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 6 (26)
Platelet count decreased (Investigations) | 4 (8)
White blood cell decreased (Investigations) | 4 (8)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT04295759/Prot_SAP_000.pdf